CLINICAL TRIAL: NCT02345317
Title: Reticular Pseudodrusen Progression Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: AltenAugenklinik
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Age-related macular degeneration (AMD) is the leading cause of irreversible blindness in industrial countries. Reticular pseudodrusen (RPD) have been recognized as an additional phenotypic characteristic frequently observed in patients with AMD. Several studies have proven that the prevalence of RPD is associated with AMD as well as a high risk of disease progression to geographic atrophy, the late form of dry AMD. The pathogenesis of RPD is yet still incompletely understood. Retrospective studies have demonstrated that the RPD affected retinal area increases over time. Potential factors influencing progression of RPD have not been intensely studied and potentially predictive markers are yet unknown. The primary objective of this study is to characterize RPD progression in more detail and to identify predictive markers of RPD progression and development of AMD late stages.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Men and women, any race, aged 60 years or older at the baseline visit
* Presence of RPD without any other type of drusen, hypo/hyperpigmentation, geographic atrophy, choroidal neovascularization
* Patient is willing to undergo ocular examinations once every 12 for up to 24 months

Exclusion Criteria:

* Presence or history of soft drusen, hypo-/hyperpigmentation, geographic atrophy or choroidal neovascularization in the study eye
* Ocular disease in the study eye that may confound assessment of the retina (e.g., diabetic retinopathy, uveitis)
* Any condition that would make adherence to the examination schedule of once every 12 months for up to 24 months difficult or unlikely, e.g., personality disorder, chronic alcoholism, Alzheimer's Disease or drug abuse

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suitable for the study will be recruited at the University of Muenster, Department of Ophthalmology
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change of reticular pseudodrusen affected retinal area to baseline | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Eter, Prof, Principal Investigator — Department of Ophthalmology, University Medical Center Muenster
Locations (1):
- Department of Ophthalmology, University Medical Center Muenster, Münster, Germany

REFERENCES:
- [Background] Alten F, Heiduschka P, Clemens CR, Eter N. Longitudinal structure/function analysis in reticular pseudodrusen. Invest Ophthalmol Vis Sci. 2014 Aug 21;55(9):6073-81. doi: 10.1167/iovs.13-13804. PMID 25146989
- [Background] Alten F, Clemens CR, Heiduschka P, Eter N. Characterisation of reticular pseudodrusen and their central target aspect in multi-spectral, confocal scanning laser ophthalmoscopy. Graefes Arch Clin Exp Ophthalmol. 2014 May;252(5):715-21. doi: 10.1007/s00417-013-2525-y. Epub 2013 Nov 26. PMID 24276561
- [Background] Alten F, Clemens CR, Heiduschka P, Eter N. Localized reticular pseudodrusen and their topographic relation to choroidal watershed zones and changes in choroidal volumes. Invest Ophthalmol Vis Sci. 2013 May 7;54(5):3250-7. doi: 10.1167/iovs.13-11923. PMID 23599330
- [Background] Alten F, Heiduschka P, Clemens CR, Eter N. Multifocal electroretinography in eyes with reticular pseudodrusen. Invest Ophthalmol Vis Sci. 2012 Sep 14;53(10):6263-70. doi: 10.1167/iovs.12-10094. PMID 22918638
- [Background] Alten F, Clemens CR, Milojcic C, Eter N. Subretinal drusenoid deposits associated with pigment epithelium detachment in age-related macular degeneration. Retina. 2012 Oct;32(9):1727-32. doi: 10.1097/IAE.0b013e3182475b03. PMID 22466490